CLINICAL TRIAL: NCT01499836
Title: Effect of Anesthetic Technique on Pain、 Recovery and Satisfaction in Women Undergoing Breast Surgery
Brief Title: Quality Study of Anesthetic Technique on Breast Cancer Surgery
Acronym: PQSAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nai Liang Li (Other)
Responsible Party: Sponsor-Investigator, Nai Liang Li, M.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110920A
Record Dates: First submitted 2011-12-10; First posted 2011-12-26 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Postoperative Pain; Quality of Recovery; Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- general anesthesia and PVB (Experimental): general anesthetics consisting of propofol, cisatracurium and fentanyl for endotracheal intubation and deaflurane for maintenance will be given. After intubation, paravertebral injections will be performed under ultrasound guidance.
  Interventions: Other: PVB
- sedation and PVB (Experimental): After sedation with midazolam and fentanyl, the patients in sedation and PVB group will receive PVB. paravertebral injections will be performed under ultrasound guidance.Intraoperative sedation will be provided with propofol titrated to moderate sedation.
  Interventions: Other: PVB
- general anesthesia (Active Comparator): general anesthetics consisting of propofol, cisatracurium and fentanyl for endotracheal intubation and deaflurane for maintenance will be given.
  Interventions: Other: PVB

INTERVENTIONS:
Other: PVB — paravertebral block

SUMMARY:
Previous studies have shown that paravertebral block (PVB) has the potential to reduce pain and side effects after breast surgery when used in addition to general anesthesia or sedation.The investigators would like to further discern the impact of GA or PVB on the postoperative QoR, pain and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a physical status between ASA I and III
* Female
* 18 - 70 years of age
* Patients able to read a newspaper in Chinese.
* Elective unilateral wide excision/simple mastectomy and SLNB/ALND
* Patient has signed an informed consent
* Without contraindication of GA or PVB
* Body mass index (BMI) less than 24 kg/m2

Exclusion Criteria:

* ASA > III
* inability to provide informed consent
* Bleeding disorders
* Contraindications to nonsteroidal anti-inflammatory drugs (NSAIDs)
* Allergy to amide-type local anesthetics or NSAIDs
* Infection at the thoracic paravertebral injection site
* Pregnancy or breast-feeding
* Severe spine or chest wall deformity
* body mass index equal to or more than 24 kg/m2
* patients with major psychosis or drug and alcohol abuse
* patients with a history of significant neurological, psychiatric, neuromuscular, cardiovascular, pulmonary, renal or hepatic disease
* Patients with significant visual impairment or other physical disability that precludes complete cooperation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
quality of recovery | postoperative 6 hour and postoperative day(POD)1

SECONDARY OUTCOMES:
adverse events | POD1
Number of patients with a technique failure of the PVB | during operation
NRS pain score | postoperative 1 hour, 6 hour, and POD1
Satisfaction | POD1

CONTACTS AND LOCATIONS:
Overall Officials: Nai Liang Li, Principal Investigator — Koo Foundation Sun Yat-Sen Cancer Center
Locations (1):
- Koo Foundation Sun Yat-Sen Cancer Center, Taipei, Taiwan, Taiwan